CLINICAL TRIAL: NCT02538354
Title: The Effect of Riboflavin Supplementation on Faecalibacterium Prausnitzii in Crohn's Disease
Brief Title: The Effect of Riboflavin in Crohn's Disease
Acronym: RISE-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. G. Dijkstra, Prof. dr. G. Dijkstra, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: METc 2014/291; Protocol ID (Other: NL-48186.042.14)
Record Dates: First submitted 2015-08-20; First posted 2015-09-02 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease
Keywords: Riboflavin (vitamin B2); Faecalibacterium prausnitzii
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riboflavin supplementation in quiescent disease (Experimental): Group 1 (n=42) will consist of patients with disease in remission (quiescent disease).
  Interventions: Dietary Supplement: Riboflavin supplementation
- Riboflavin supplementation in active disease (Experimental): Group 2 (n=42) will consist of patients with active disease.
  Interventions: Dietary Supplement: Riboflavin supplementation

INTERVENTIONS:
Dietary Supplement: Riboflavin supplementation — Supplementation of the normal diet with 1 capsule of 100 mg riboflavin (vitamin B2) during three weeks
  Other Names: vitamin B2 supplementation

SUMMARY:
This study will evaluate if suppelementation of the diet with riboflavin in Crohn's disease patients will result in an increase in the amount of F. prausnitzii.

DETAILED DESCRIPTION:
Rationale Recent studies show that in patients with Inflammatory Bowel Disease (IBD) a dysbiosis exists in the composition of the intestinal microbiota. In particular, the potentially pathogenic bacterium Escherichia coli (E. coli) is often more abundant in the bowel of IBD patients, and the anaerobic commensal Faecalibacterium prausnitzii (F. prausnitzii) is often reduced. This last mentioned bacteria is known to be abundant in the intestine of healthy individuals. It is known to produce butyrate, which stimulates the intestinal epithelium, and to secrete anti-inflammatory substances.

Riboflavin - also known as vitamin B2 - is required for a wide variety of cellular processes and has an important role in maintaining health in humans. In a pilot intervention with healthy volunteers it is shown that a riboflavin supplement increases the number of F. prausnitzii and results in a higher production of butyrate. In Crohn's disease patients, it is known that the amount of F. prausnitzii in the intestine is generally low. Furthermore, it is known that there is an association between the number of F. prausnitzii bacteria and the length of disease in remission.

This study will evaluate if supplementation of the diet with riboflavin in Crohn's disease patients will result in a similar increase in the amount of F. prausnitzii as in healthy volunteers. In this patient group, an increase in the number of F. prausnitzii bacteria in the bowel may result in a more favourable disease course. This will be assessed with faeces calprotectin and two questionnaires. Additionally the investigators will assess if there is any modulation by riboflavin on the other intestinal bacteria, short chain fatty acids (SCFAs) (such as butyrate), and the pH of the faeces. Finally, the effect of the riboflavin on the permeability of the gut will be evaluated with a Chroom-EDTA test, and a number of different biomarkers of permeability.

Hypothesis The hypothesis is that in Crohn's disease patients, supplementation of the diet with riboflavin results in an increase in the amount of F. prausnitzii, changes in microbial composition, increased fatty acid production, an increase in pH and a reduction of intestinal permeability. These changes might result in a more favourable disease course with less exacerbations.

Study design Prospective clinical study.

Study population and sample size In total 84 Crohn's disease patients will be included in this study, divided into two groups. Group 1 (n=42) will consist of patients with disease in remission (quiescent disease); group 2 (n=42) will consist of patients with active disease. In this study an adaptive design will be used. First 12 patients in the disease in remission group will be analysed. The methods of analysis and safety aspects will be taken into account.

Intervention Supplementation of the normal diet with 1 capsule of 100 mg riboflavin (vitamin B2) during three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease patients
* Age 18-65 years
* Concomitant medication for Crohn's disease is allowed in all groups

Exclusion Criteria:

* Swallowing disorders
* Pregnancy and lactation
* Use of antibiotic drugs, probiotics (i.e.Yakult, Vifit, Activia etc) or specific prebiotic supplements in the 3 weeks prior to the riboflavin intervention
* Use of Methotrexate drugs
* Colonoscopy and colon cleansing in last 3 months
* Use of a vitamin B2 supplement, or multivitamin complexes containing vitamin B (i.e. vitamin B-complex) in the 3 weeks prior to the riboflavin intervention
* Severe Crohn's disease (HBI > 12)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Sartor RB. Microbial influences in inflammatory bowel diseases. Gastroenterology. 2008 Feb;134(2):577-94. doi: 10.1053/j.gastro.2007.11.059. PMID 18242222
- [Background] Sokol H, Pigneur B, Watterlot L, Lakhdari O, Bermudez-Humaran LG, Gratadoux JJ, Blugeon S, Bridonneau C, Furet JP, Corthier G, Grangette C, Vasquez N, Pochart P, Trugnan G, Thomas G, Blottiere HM, Dore J, Marteau P, Seksik P, Langella P. Faecalibacterium prausnitzii is an anti-inflammatory commensal bacterium identified by gut microbiota analysis of Crohn disease patients. Proc Natl Acad Sci U S A. 2008 Oct 28;105(43):16731-6. doi: 10.1073/pnas.0804812105. Epub 2008 Oct 20. PMID 18936492
- [Background] Fujimoto T, Imaeda H, Takahashi K, Kasumi E, Bamba S, Fujiyama Y, Andoh A. Decreased abundance of Faecalibacterium prausnitzii in the gut microbiota of Crohn's disease. J Gastroenterol Hepatol. 2013 Apr;28(4):613-9. doi: 10.1111/jgh.12073. PMID 23216550
- [Background] Willing B, Halfvarson J, Dicksved J, Rosenquist M, Jarnerot G, Engstrand L, Tysk C, Jansson JK. Twin studies reveal specific imbalances in the mucosa-associated microbiota of patients with ileal Crohn's disease. Inflamm Bowel Dis. 2009 May;15(5):653-60. doi: 10.1002/ibd.20783. PMID 19023901
- [Background] Sokol H, Seksik P, Furet JP, Firmesse O, Nion-Larmurier I, Beaugerie L, Cosnes J, Corthier G, Marteau P, Dore J. Low counts of Faecalibacterium prausnitzii in colitis microbiota. Inflamm Bowel Dis. 2009 Aug;15(8):1183-9. doi: 10.1002/ibd.20903. PMID 19235886
- [Background] Miquel S, Martin R, Rossi O, Bermudez-Humaran LG, Chatel JM, Sokol H, Thomas M, Wells JM, Langella P. Faecalibacterium prausnitzii and human intestinal health. Curr Opin Microbiol. 2013 Jun;16(3):255-61. doi: 10.1016/j.mib.2013.06.003. Epub 2013 Jul 3. PMID 23831042
- [Background] Louis P, Flint HJ. Diversity, metabolism and microbial ecology of butyrate-producing bacteria from the human large intestine. FEMS Microbiol Lett. 2009 May;294(1):1-8. doi: 10.1111/j.1574-6968.2009.01514.x. Epub 2009 Feb 13. PMID 19222573
- [Background] Khan MT, Duncan SH, Stams AJ, van Dijl JM, Flint HJ, Harmsen HJ. The gut anaerobe Faecalibacterium prausnitzii uses an extracellular electron shuttle to grow at oxic-anoxic interphases. ISME J. 2012 Aug;6(8):1578-85. doi: 10.1038/ismej.2012.5. Epub 2012 Feb 23. PMID 22357539
- [Background] Swidsinski A, Loening-Baucke V, Vaneechoutte M, Doerffel Y. Active Crohn's disease and ulcerative colitis can be specifically diagnosed and monitored based on the biostructure of the fecal flora. Inflamm Bowel Dis. 2008 Feb;14(2):147-61. doi: 10.1002/ibd.20330. PMID 18050295

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riboflavin Supplementation in Quiescent Disease | Riboflavin Supplementation in Active Disease
Started | 40 | 30
Completed | 40 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riboflavin Supplementation in Quiescent Disease | Riboflavin Supplementation in Active Disease | Total
Number analyzed (Participants) | 40 | 30 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.6) | 38.8 (13.6) | 41.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 19 | 48
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 40 | 30 | 70

OUTCOME MEASURES:

1. Primary Outcome: F. Prausnitzii (FISH Analysis).
Description: The faeces is collected at different time points before and after riboflavin supplementation. To investigate the effect of a riboflavin supplement on the number of F. prausnitzii bacteria in the faeces of active and quiescent Crohn's disease patients.
Time Frame: Different time points up to 6 weeks from start study: Day0, Day7, Day28
Measure: Median (Inter-Quartile Range); unit: Relative FISH counts from total bacteria
Arm/Group | Riboflavin Supplementation in Quiescent Disease | Riboflavin Supplementation in Active Disease
Number analyzed (Participants) | 40 | 30
Relative FISH counts from total bacteria
  T0 (Mean of Day 0 and Day 7 combined) | 4.53 [0.00 to 12.77] | 5.07 [0.00 to 14.03]
  T3 (Day 28) | 6.19 [0.00 to 13.10] | 5.46 [0.00 to 11.98]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: No adverse events observed in this study
Arm/Group | Riboflavin Supplementation in Quiescent Disease | Riboflavin Supplementation in Active Disease
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/30
Other Adverse Events (participants affected / at risk) | 0/40 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02538354/Prot_SAP_000.pdf